CLINICAL TRIAL: NCT00030706
Title: Phase II Study Of Epothilone B Analogue BMS-247550 In Relapse And/Or Refractory Stage III Or IV Ovarian Epithelial Cancer, Following Front-Line Treatment With Platinum Plus Taxane-Based Chemotherapy
Brief Title: Ixabepilone in Treating Patients With Relapsed and/or Refractory Stage III or Stage IV Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069190; P30CA013330 (NIH); AECM-3632; MCC-12602; NCI-3632
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — ixabepilone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ixabepilone in treating patients who have relapsed and/or refractory stage III or stage IV ovarian epithelial cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of ixabepilone, in terms of clinical response and progression-free survival, in patients with relapsed and/or refractory stage III or IV ovarian epithelial or primary peritoneal cancer.
* Determine the nature and degree of toxicity of this drug in these patients.

Secondary

* Correlate pre-ixabepilone survivin mRNA and protein levels in patient-derived ovarian cancer cells with quality of response (i.e., at least partial response vs no response).
* Correlate CYP3A4 (3A4*1B), 3A5 (3A5*1), and 3A7 (ER6 p variation) allelic polymorphisms with parent drug kinetic parameters, toxicity, and efficacy of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive ixabepilone IV over 1 hour once weekly on weeks 1-3. Treatment repeats every 4 weeks for a total of 3 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage III or IV ovarian epithelial cancer or primary peritoneal carcinoma

  * Recurrent or refractory disease

    * Previously treated with 1, and only 1, prior chemotherapy regimen containing carboplatin, cisplatin, or another organoplatinum compound and paclitaxel or docetaxel
    * Initial treatment may include high-dose, consolidation, or extended therapy administered after surgical or non-surgical assessment
* Bidimensionally measurable disease by physical exam, CT scan, or MRI

  * Ascites and pleural effusions are not measurable disease
  * No prior irradiation to indicator lesions

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No prior bleeding disorder or unexplained bleeding

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Other

* No active infection requiring antibiotics
* No grade 2 or greater neuropathy (sensory and motor)
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No prior recurrent grade 2 or greater hypersensitivity reactions to Cremophor EL, docetaxel, or paclitaxel
* No other medical condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior biologic or immunologic therapy for ovarian epithelial or primary peritoneal carcinoma

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered
* No prior ixabepilone
* No prior cytotoxic chemotherapy (including retreatment with initial chemotherapy regimens) for recurrent or persistent ovarian epithelial or primary peritoneal carcinoma

Endocrine therapy

* At least 1 week since prior hormonal therapy for ovarian epithelial or primary peritoneal carcinoma
* Concurrent hormonal replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to a site of measurable disease used on study
* No prior radiotherapy to more than 25% of bone marrow

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* At least 3 weeks since other prior therapies for ovarian epithelial or primary peritoneal carcinoma
* No prior cancer treatment for other invasive malignancies that would preclude study participation
* No concurrent heparin or other anticoagulants
* No concurrent Hypericum perforatum (St. John's wort) or any product containing this compound

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11 (Actual); Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical remission | up to 12-months post-treatment
  number of participants experience clinical remission will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Goldberg, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York, United States